CLINICAL TRIAL: NCT04239924
Title: Community Paramedic Coaching Program for Caregivers and People With Dementia (CP3D)
Brief Title: Community Paramedic Coaching Program for Caregivers and People With Dementia
Acronym: CP3D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-1218; A534100 (Other: UW Madison); SMPH/EMERG MED (Other: UW Madison); K24AG054560 (NIH); Protocol Version 1/20/2021 (Other: UW Madison)
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Dementia
Keywords: Community Care; Coaching; Paramedic; Caregivers
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Paramedic Coaching (Experimental): The intervention is an adaptation of the evidence-based REACH program
  Interventions: Behavioral: Paramedic Coaching

INTERVENTIONS:
Behavioral: Paramedic Coaching — The intervention is an adaptation of the evidence-based REACH program, specific coaching content is delivered by paramedics in 1-2 hour in-home sessions and over the phone throughout a 12-month period.

SUMMARY:
This pilot study is designed to evaluate the potential effectiveness of the implementation strategy and intervention delivery model of a community paramedic coaching program for caregivers of persons with dementia, in direct coordination with the participant and caregiver's primary health care team. Specifically, the acceptability, appropriateness, and feasibility of the program will be assessed, collecting data from all implementation stakeholders at baseline, 13 weeks, 25 weeks, and post-intervention (~50 weeks) using quantitative survey instruments and qualitative interviews.

DETAILED DESCRIPTION:
The intervention is an adaptation of the evidence-based REACH program (Resources Enhancing Alzheimer's Caregiver Health), designed for and validated in multiple settings to give education, tools, and support to informal caregivers of people with dementia, delivered through a series of at-home visits (minimum of 9 in-person and 3 phone sessions) conducted by trained and certified coaches over 6-12 months. The content of the coaching visits will follow the REACH program protocol, with materials customized with information about local community resources (e.g., Dane County).

Coach/administrator training for delivery of the REACH intervention will be conducted by master trainers from the Rosalynn Carter Institute (RCI) for Caregiving, a department of Georgia Southwestern State University, who administers, certifies, and provides oversight for REACH sites nationally (https://www.rosalynncarter.org/programs/rci-reach/). For the purposes of this pilot study, the investigators have coordinated with RCI to extend delivery of REACH content over a 12-month period, with home visits occurring more frequently at the beginning and spreading further apart towards the end, and additional phone "REVIEW" sessions between home-visits.

Each home visit covers specific coaching content, building on strategies and behaviors covered in prior sessions. The program includes flexibility to allow coaches to adapt the timing/delivery of content to attend to the needs of the caregiver (e.g., answering questions about previously-covered topics, covering topics from a future visit to help coach a caregiver through an emergent dementia-related issue). Sessions typically last 1-2 hours. Following each visit, the coach completes a fidelity checklist and writes client progress notes as per the REACH protocol.

This pilot adapts prior REACH implementations in two main ways: (1) intervention coaches will be community paramedics with advanced medical training, rather than social workers (or other non-medical social service personnel), and (2) the program will be formally coordinated with the participant and caregiver's primary care practice, allowing for care coordination and information sharing between participants, coaches, and clinic staff/providers. Participants will also have the ability to share information about their use of community dementia care resources (e.g., social services, transportation, senior center case management, dementia caregiver support groups, dementia-related educational programming, respite) with coaches so they can communicate necessary information to the clinic for possible inclusion in the participant's Electronic Health Record (EHR) (as per the clinic's determination), facilitate care coordination, and help keep the participant's care plan up to date. Paramedic coaches will be utilizing their medical knowledge, but not providing any direct medical care.

This pilot study also differs from prior REACH trials in that outcome measures include health care and emergency services utilization, particularly related to the occurrence of acute medical and behavioral problems, as well as perceptions of health care quality, in addition to caregiver psycho-socio-emotional measures (already included in the standard REACH assessment package).

The study will employ a stepped design using a rapid-cycle evaluation approach. Three cohorts of 4-5 patient-caregiver dyads each will start the intervention at staggered intervals. Within each cohort, a new dyad will begin the program approximately every two weeks, with an approximate four week gap between each cohort for feedback collection and program iteration. Real-time feedback obtained from multiple intervention stakeholders (caregivers, persons with dementia, coaches, clinical staff/providers - up to 10 enrolled) will be used to iteratively improve intervention delivery and program implementation for the next, all while the first group continues the pilot. In this way, problems can be identified and solutions generated, with enough time to adapt the program and evaluate revisions. Staggering participant start dates allows for multiple rapid-cycle iterations within a single pilot study.

NOTE: While COVID-19 restrictions are in place, all feedback interviews will take place by telephone or WebEx videoconferencing, beginning 17 March 2020.

ELIGIBILITY:
Patient Inclusion Criteria:

* Diagnosis or indication in medical record of mild to moderate dementia (any subtype)
* English speaking
* Community-dwelling (independent and assisted living acceptable)
* Living with their primary informal caregiver
* Patient of a UW Health primary care provider affiliated with and participating in the study

Patient Exclusion Criteria:

* Receiving intensive care management services
* Receiving aggressive care for another condition (e.g., chemotherapy for cancer, surgery planned for problem)
* In isolation due to contagious illness
* Enrolled in home hospice
* Currently incarcerated, in police custody, or ward of the state
* Legally blind or deaf (unable to hear or see even with assistive devices)
* Lacks decisional capacity and no available legally authorized representative (LAR) to provide consent
* Patient refuses enrollment

Caregiver Inclusion Criteria:

* Adult informal caregiver (≥18 years old) of a person eligible for this study (determination based upon caregiver self-identification).
* Lives in the same household (primary residence) as the patient with dementia.
* Has a working telephone
* English speaking
* UW Health primary care provider

Caregiver Exclusion Criteria:

* Unable to participate in the program as defined
* Employed by a professional/private agency to provide care to the care recipient (i.e., professional caregiver, not an informal caregiver)
* Has a diagnosis of dementia or cognitive impairment causing functional impairment
* In isolation due to contagious illness
* Legally blind or deaf (unable to hear or see even with assistive devices)
* Refuses enrollment

Stakeholder Inclusion Criteria:

* Involved in the implementation study activities in related to the intervention, either as a clinician, member of the UW Health staff, paramedic coach, or social service provider.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manish N Shah, MD, MPH, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 participant enrolled are 10 caregivers and 10 patients with dementia
Groups:
- Paramedic Coaching of Caregivers: The intervention is an adaptation of the evidence-based REACH program
  Paramedic Coaching: The intervention is an adaptation of the evidence-based REACH program, specific coaching content is delivered by paramedics in 1-2 hour in-home sessions and over the phone throughout a 12-month period.
Period: Overall Study
Arm/Group | Paramedic Coaching of Caregivers
Started | 20
Caregivers | 10
Patient With Dementia | 10
Completed | 18
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Paramedic Coaching
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 77.1 [51 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Visits to the Emergency Department by the Person With Dementia
Description: As determined by abstracting the medical records, the investigators are testing the hypothesis that the number of visits to the Emergency Department is lower than commonly reported in the literature for persons with dementia.
Time Frame: up to 24 months
Measure: Number; unit: visits to the Emergency Department
Arm/Group | Paramedic Coaching
Number analyzed (Participants) | 10
visits to the Emergency Department | 15

2. Primary Outcome: Number of Visits to the Emergency Department by the Caregiver of the Person With Dementia
Description: As determined by abstracting the medical records, the investigators are testing the hypothesis that the number of visits to the Emergency Department is lower than commonly reported in the literature for average older adults.
Time Frame: up to 24 months
Measure: Number; unit: visits to the Emergency Department
Arm/Group | Paramedic Coaching
Number analyzed (Participants) | 10
visits to the Emergency Department | 1

3. Primary Outcome: Feasibility: Proportion of Coaching Phone Calls Completed
Description: The intervention will be deemed feasible if at least 75% of the intended coaching phone calls are completed. The minimum number of coaching calls is 3, additional calls will be scheduled opposite weeks of home visits as needed.
Time Frame: up to 12 months
Population: The coaching phone calls are relevant to and only conducted with caregivers, which makes up for 10 of our 20 participants.
Measure: Number; unit: Number of Phone Calls Completed
Units Other Than Participants: Number of Phone Calls Made
Arm/Group | Paramedic Coaching
Number analyzed (Participants) | 10
Number analyzed (Number of Phone Calls Made) | 30
Number of Phone Calls Completed | 27

4. Primary Outcome: Feasibility: Proportion of Coaching Home Visits Completed
Description: The intervention will be deemed feasible if at least 75% of the intended home visits are completed. The minimum number of intended home visits is 9.
Time Frame: up to 12 months
Population: as for outcome 3
Measure: Number; unit: number of completed coaching visits
Units Other Than Participants: Number of Home Visits Planned
Arm/Group | Paramedic Coaching
Number analyzed (Participants) | 10
Number analyzed (Number of Home Visits Planned) | 90
number of completed coaching visits | 82

5. Secondary Outcome: Change in Zarit Burden Interview (ZBI-12) Score
Description: The Zarit Burden Interview measures caregiver burden. This is a 12-item survey with a total possible range of scores from 0-48, where higher scores indicate increased burden. The investigators hypothesize the score will decrease as a result of the intervention.
Time Frame: First home visit (~ week 1), week 13, week 25, and last home visit (~up to week 50)
Population: This interview is relevant to and only conducted on caregivers, which makes up for 10 of our 20 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Paramedic Coaching of Caregivers
Number analyzed (Participants) | 10
score on a scale
  First home visit: number analyzed (Participants) | 8
  First home visit | 13 (9.7)
  Week 13: number analyzed (Participants) | 8
  Week 13 | 18.5 (11.7)
  Week 25: number analyzed (Participants) | 8
  Week 25 | 15.75 (7.8)
  Week 50: number analyzed (Participants) | 1
  Week 50 | 19 (NA) — Unable to obtain standard deviation with sample size of 1. By week 50, we were only able to obtain 1 participant's feedback.

6. Secondary Outcome: Change in Generalized Anxiety Disorder (GAD-7) Score
Description: The GAD-7 is a 7-item survey that measures anxiety symptom severity. The total possible range of scores is 0-21, where higher scores indicate increased symptom severity. The investigators hypothesize the score will decrease as a result of the intervention.
Time Frame: Baseline, week 13, week 25, week 50
Population: This interview is relevant to and only conducted on caregivers, which makes up for 10 of our 20 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Paramedic Coaching of Caregivers
Number analyzed (Participants) | 10
score on a scale
  Baseline | 7.7 (4.7)
  Week 13: number analyzed (Participants) | 8
  Week 13 | 5.5 (3.3)
  Week 25: number analyzed (Participants) | 8
  Week 25 | 5.4 (3.0)
  Week 50: number analyzed (Participants) | 1
  Week 50 | 4 (NA) — Unable to obtain standard deviation with sample size of 1. By week 50, we were only able to obtain 1 participant's feedback.

7. Secondary Outcome: Change in Center for Epidemiologic Studies Depression Scale (CESD-10)
Description: The CESD-10 is a general measure of depression frequently used in caregiver studies. It is a 10-item survey with a total possible range of scores of 0-30 where higher scores indicate increased depression. The investigators hypothesize the score will decrease as a result of the intervention.
Time Frame: First home visit (~ week 1), week 13, week 25, and last home visit (~up to week 50)
Population: This interview is relevant to and only conducted on caregivers, which makes up for 10 of our 20 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Paramedic Coaching of Caregivers
Number analyzed (Participants) | 10
score on a scale
  First home visit: number analyzed (Participants) | 9
  First home visit | 7.7 (5.7)
  Week 13: number analyzed (Participants) | 8
  Week 13 | 8.4 (4.5)
  Week 25: number analyzed (Participants) | 9
  Week 25 | 7.3 (5.4)
  Week 50: number analyzed (Participants) | 1
  Week 50 | 10 (NA) — Unable to obtain standard deviation with sample size of 1. By week 50, we were only able to obtain 1 participant's feedback.

8. Secondary Outcome: Change in Revised Caregiving Satisfaction Scale (RCSS)
Description: The RCSS is a 6-item survey used to measure the positive aspects of caring. The range of total possible scores is 6-30 where higher scores indicate increased caregiver satisfaction. The investigators hypothesize the score will increase as a result of the intervention.
Time Frame: Baseline, week 13, week 25, week 50
Population: This interview is relevant to and only conducted on caregivers, which makes up for 10 of our 20 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Paramedic Coaching of Caregivers
Number analyzed (Participants) | 10
score on a scale
  Baseline: number analyzed (Participants) | 9
  Baseline | 24.1 (3.6)
  Week 13: number analyzed (Participants) | 8
  Week 13 | 20.5 (4.1)
  Week 25: number analyzed (Participants) | 8
  Week 25 | 22 (4.9)
  Week 50: number analyzed (Participants) | 1
  Week 50 | 24 (NA) — Unable to obtain standard deviation with sample size of 1. By week 50, we were only able to obtain 1 participant's feedback.

9. Secondary Outcome: Change in Revised Scale for Caregiving Self-Efficacy
Description: The revised scale for caregiving self-efficacy measures three domains: obtaining respite, responding to disruptive patient behaviors, and controlling upsetting thoughts. It is a 15-item scale with a total possible range of scores between 0-100, where higher scores are better. The investigators hypothesize the score will increase as a result of the intervention.
Time Frame: First home visit (~ week 1) and last home visit (~up to week 50)
Population: This interview is relevant to and only conducted on caregivers, which makes up for 10 of our 20 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Paramedic Coaching of Caregivers
Number analyzed (Participants) | 10
score on a scale
  Obtaining Respite - first home visit | 65.8 (28.2)
  Obtaining Respite - last home visit | 71.6 (18.9)
  Responding to Disruptive Behavior - first home visit | 70.4 (11.8)
  Responding to Disruptive Behavior - last home visit | 77.6 (12.7)
  Controlling Upsetting Thoughts - first home visit | 76.22 (12.7)
  Controlling Upsetting Thoughts - last home visit | 78.4 (10.6)

10. Secondary Outcome: Change in Work-Family Conflict Scale (WFC)
Description: WFC is measured for the caregiver. It is a 6-item survey with a total possible range of scores between 6-30 with higher scores indicating lesser work-family conflict. The investigators hypothesize the score will increase as a result of the intervention.
Time Frame: First home visit (~ week 1) and last home visit (~up to week 50)
Population: Survey only relevant to caregivers who are working. Unable to obtain participant feedback for last home visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Paramedic Coaching of Caregivers
Number analyzed (Participants) | 4
score on a scale
  First Home Visit | 15 (3.9)
  Last Home Visit: number analyzed (Participants) | 0

11. Secondary Outcome: Change in Caregiver Quality of Life (C-DEMQOL) Score
Description: C-DEMQOL is measured for the caregiver. The investigators will be asking 18 of the questions from the scale to understand the quality of life the caregivers experience. Scores can range from 18-90, with a higher score reflecting a higher quality of life.
Time Frame: First home visit (~ week 1), week 13, week 25, and last home visit (~up to week 50)
Population: This interview is relevant to and only conducted on caregivers, which makes up for 10 of our 20 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Paramedic Coaching of Caregivers
Number analyzed (Participants) | 10
score on a scale
  First home visit: number analyzed (Participants) | 9
  First home visit | 20.4 (4.4)
  Week 13: number analyzed (Participants) | 8
  Week 13 | 20.4 (4.4)
  Week 25: number analyzed (Participants) | 8
  Week 25 | 20.5 (3.7)
  Week 50: number analyzed (Participants) | 3
  Week 50 | 19.5 (4.0)

12. Secondary Outcome: Change in Knowledge of Dementia (DKAS) Score
Description: DKAS is measured for the caregiver. It is a 25 item true-false survey of facts about dementia. Scoring is by measuring the proportion of questions answered correctly. The range for score values is 0 to 50, the higher the score the better the outcome (a.k.a. the more knowledgeable about dementia).
Time Frame: First home visit (~ week 1) and week 13
Population: This interview is relevant to and only conducted on caregivers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Paramedic Coaching of Caregivers
Number analyzed (Participants) | 8
score on a scale
  First home visit | 34.3 (3.5)
  Week 13 | 35 (5.6)

13. Secondary Outcome: Clinic Utilization by Persons With Dementia
Description: As determined by abstracting the medical records, the investigators are characterizing the number of contacts with outpatient clinics for persons with dementia.
Time Frame: up to 24 months
Population: No data was collected. As the outcomes were not relevant to the primary goal of the project, medical records were not abstracted for this data due to study staff changes and time constraints.
Arm/Group | Paramedic Coaching of Caregivers
Number analyzed (Participants) | 0

14. Secondary Outcome: Clinic Utilization by Caregivers of Persons With Dementia
Description: As determined by abstracting the medical records, the investigators are characterizing the number of contacts with outpatient clinics for caregivers of persons with dementia.
Time Frame: up to 24 months
Population: as for outcome 13
Arm/Group | Paramedic Coaching of Caregivers
Number analyzed (Participants) | 0

15. Secondary Outcome: Change in Caregiver Perceptions About Communication With Clinical Team Members (CAPACITY) Measure
Description: Assesses caregivers perception of communication with health care team and extent to which the team considers their capacity and preferences in decision making. This measure consists of 12 questions, with scores ranging from 12-60, where higher scores indicate increased communication with the health care team.
Time Frame: First home visit (~ week 1) and week 13
Population: This interview is relevant to and only conducted on caregivers, which makes up for 10 of our 20 participants.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Paramedic Coaching of Caregivers
Number analyzed (Participants) | 10
score on a scale
  First home visit | 32.3 (8.8)
  Week 13 | 36.6 (2.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time a participant was enrolled to 6 months after the completion of their participation. Typically, 1 year and 6 months.
Description: Adverse events for caregivers and for patients with dementia were not monitored/assessed separately.
Arm/Group | Paramedic Coaching
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 7/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paramedic Coaching (N=20)
Serious Adverse Events (Vascular disorders) | 1 (2) — Pt presented w/ stroke symptoms of LE weakness. MRI showed acute right thalamic infarct & vascular imaging showed no flow limiting stenosis of carotids. Pt given aspirin, statin, antihypertensives. Pt d/c to f/u w/ stroke clinic, & rec'd home health
Serious Adverse Event (Vascular disorders) | 1 (1) — Pt presented to ED c/o 2 weeks worsening chest pain w/ SOB. Pt HTN in ED. CXR, Trops and ECG WNL. CT shows no PE. After admission pt able to complete walking desaturation test, HTN decreased. Pt d/c w/ instructions to f/u w/ PCP.
Serious Adverse Event (General disorders) | 1 (1) — Pt presented to ED c/o worsening LE weakness. Pt admitted after elevated trop-NSTEMI type 2 demand. Cardiology placed pt on heparin infusion for 48 hrs. Pt stable, LLL pneumonia resolved with IV abx. D/c to SNF for PT/OT therapy & f/u w/ PCP & Cardio
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paramedic Coaching (N=20)
ED Use (Renal and urinary disorders) | 1 (3) — 3 visits to ED for Urinary Catheter Problem within 1 week
ED Use (Vascular disorders) | 1 (1) — Pt presented to ED with Dizziness
ED Use (Nervous system disorders) | 1 (1) — Pt presented to ED with Altered Mental Status
ED Use (Vascular disorders) | 1 (1) — Pt presented to ED with Hypertension
ED Use (Vascular disorders) | 1 (1) — Pt presented to ED with Chest Pain
ED Use (Gastrointestinal disorders) | 1 (2) — Pt presented to ED with Abdominal Pain twice in one week
ED Use (Injury, poisoning and procedural complications) | 1 (1) — Pt presented to ED with Fall
ED Use (Vascular disorders) | 1 (1) — Pt presented to ED with Weakness
ED Use (General disorders) | 1 (1) — Pt presented to ED with Leg Problem

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT04239924/Prot_SAP_000.pdf
  • Informed Consent Form: Caregiver Informed Consent Form (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT04239924/ICF_001.pdf
  • Informed Consent Form: Patient with Dementia Informed Consent Form (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT04239924/ICF_002.pdf